CLINICAL TRIAL: NCT04630899
Title: Comparison of Passive and Active Joint Mobilization for Chronic Ankle Instability: a Randomized Controlled Trial
Brief Title: Comparison of Passive and Active Joint Mobilization for Chronic Ankle Instability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sahmyook University (Other)
Responsible Party: Principal Investigator, Hyunjoong Kim, Principal Investigator, Sahmyook University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P01-202105-11-003
Record Dates: First submitted 2020-11-08; First posted 2020-11-16 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Musculoskeletal Manipulations; Chronic Instability of Joint; Ankle Joint

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active Joint Mobilization (Experimental)
  Interventions: Other: Active joint mobilization
- Passive Joint Mobilization (Experimental)
  Interventions: Other: Passive joint mobilization

INTERVENTIONS:
Other: Active joint mobilization — The participants bend his knees in a prone position. The physical therapist holds the medial malleolus with one hand and the lateral malleolus with the other. At the same time, the physical therapist touches the participant's soles to the sternum area and presses them in the dorsal direction. At this time, medial malleolus glides anterior and lateral malleolus glides posterior. The first procedure is to passively recognize movement. The second procedure is accompanied by active movement of the participant.
  Arms: Active Joint Mobilization
Other: Passive joint mobilization — PJM uses Maitland's Mobilization method, grade III (high amplitude in the end range of the joint and 1 second vibration in the middle range through linear motion in which tissue resistance is felt). The participant is in a supine position, and the physical therapist holds the talus with one hand and the tibia with the other hand, and performs joint mobilization in the posterior direction with the hand holding the talus.
  Arms: Passive Joint Mobilization

SUMMARY:
The features of CAI were confirmed through studies that 64% to 77% had extra-articular conditions mainly related to calf tendon disorder. In addition, joints are laxity, sensory motors are deficient, and the range of dorsi flexion is decreased. this study is to investigate the effects of active joint mobilization(AJM) under weight-bearing conditions to stimulate various proprioceptors for CAI with deficiency in sensorimotor and postural control.

ELIGIBILITY:
Inclusion Criteria:

* First ankle sprain one year before clinical trial
* A score of less than 24 on the Cumberland Ankle Instability Tool (CAIT)
* No ankle sprains occurred within 4 weeks of starting the test
* Two or more more ankle sprains in the past month

Exclusion Criteria:

* If you have a history of lower extremity surgery
* In case of receiving treatment for the affected ankle within 1 month
* If you have a psychological problem

Ages: 19 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2021-09-30 (Actual); Primary Completion 2021-12-10 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Ankle instability | 4 weeks
  Consists of 9 questions, 3 to 0 points for 5 questions, 4 to 0 points for 2 questions, 5 to 0 points for 1 question, and 2 to 0 points for another question. A total score of 30 points is the highest, 28 points or more are stable ankle joints, and 24 points or less are unstable ankle joints. The higher the score, the closer to normal, and the lower the score, the lower the stability.
Range of motion | 4 weeks
  Measured based on the accelerometer sensor built into the mobile phone with a clinometer app. After fixing the mobile phone on the participant's sole, press "0 clear" to calibrate it to the initial value. The physical therapist asks the participant to "flex the foot in the dorsal direction " Measure a total of 2 times and record it as an average value.

CONTACTS AND LOCATIONS:
Locations (1):
- Gwangju Health University, Gwangju, South Korea